CLINICAL TRIAL: NCT04427657
Title: Adipose Microfragmented Autologous Tissue for the Treatment of Knee Osteoarthritis
Brief Title: Use of Lipogems for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LipoOA
Record Dates: First submitted 2020-04-22; First posted 2020-06-11 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Active Comparator): 39 patients with knee osteoarthritis undergoing arthroscopic debridement
  Interventions: Procedure: arthroscopic debridment
- Cases (Experimental): 39 patients with knee osteoarthritis undergoing arthroscopic debridement surgery + intrarticular injection of autologous microfragmented lipoaspirate tissue (Lipogems®).
  Interventions: Procedure: autologous microfragmented lipoaspirate tissue (Lipogems®).

INTERVENTIONS:
Procedure: autologous microfragmented lipoaspirate tissue (Lipogems®). — patient in supine position. A double contemporary operating fields is made under sedation. During arthroscopic debridement is made an injection of local anesthetic at the dermal level with a subcutaneous infiltration of Klein solution. The plastic surgeon wait for about 5 minutes for vasoconstriction and then start with liposuction of about 60 ml of adipose tissue. Then lipoaspirate was processed with Lipogems® technique that consist in a mechanical fragmentation, physiological washing and filter passage of the lipoaspirate. A volume of 8-9 ml of microfragmented adipose tissue was injected intra-articulary after arthroscopic debridement.
  Arms: Cases
Procedure: arthroscopic debridment — patient in supine position. Under sedation is perform an arthroscopic debridement
  Arms: Controls

SUMMARY:
Lipogems system consist in the use of a monouse kit for liposuction, processing and administration of adipose tissue. The use of the final product (microfragmented adipose tissue,not expanded) shoud promote the natural joint homeostasis, associated with a clinical improvement

DETAILED DESCRIPTION:
The Objectiveof the study is to analyse the therapeutic role of microfragmented autologous tissue for the treatment of the knee osteoarthritis (OA).

Main purpose: Symptomatic and functional evaluation at 6 months by comparison of the Knee Injury and Osteoarthritis Outcome Score(KOOS) recorded between two groups (6±1 months) undergoing arthroscopic debridement ± injection of autologous microfragmented lipoaspirate tissue (Lipogems®).

Secondary Purposes: Evaluation of possible radiological changes pre-operative and after 6±1 months by means of MagneticResonanceImage analysis. Symptomatic and functional evaluation at 6±1 months by means of VisualAnalogueScale, KneeSocietyScore, Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC). Reduction of anti-inflammatory drugs (pre-intervention versus 6±1 months). Evaluation "quality-adjusted life years" (QUALY) in relation to the questionnaire SatisfactioForm-12 (pre-intervention vs 6±1 months). Check for any adverse effects directly related to the use of micro-fragmented adipose tissue. Changes in serum levels of biomarkers related to OA (CollagenType II C-Telopeptide (CTX-II), collagen type III N-propeptide (PIIINP)) will be evaluated (pre-intervention vs 6±1 months).

The study is an interventional, prospective, randomized, controlled trial. Controls: n = 39 patients with knee osteoarthritis undergoing arthroscopic debridement. Cases: n = 39 patients with knee osteoarthritis undergoing arthroscopic debridement surgery + intrarticular injection of autologous microfragmented lipoaspirate tissue (Lipogems®).

Surgical technique: patient in supine position. A double contemporary operating fields is made under sedation. During arthroscopic debridement is made an injection of local anesthetic at the dermal level with a subcutaneous infiltration of Klein solution. The plastic surgeon wait for about 5 minutes for vasoconstriction and then start with liposuction of about 60 ml of adipose tissue. Then lipoaspirate was processed with Lipogems® technique that consist in a mechanical fragmentation, physiological washing and filter passage of the lipoaspirate. A volume of 8-9 ml of microfragmented adipose tissue was injected intra-articulary after arthroscopic debridement.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis grade III e IV Kellgren-Lawrence,
* age between 45 and 75,
* pain ≥ 6 VAS scale,
* no ligamentous instability,axial deviation less than 10°
* BMI between 18 and 30,
* International Normalized Ratio (INR) < 1.5

Exclusion Criteria:

* previous traumatic lesion (tibial fracture, osteothomy) of the knee
* osteonecrosis
* meniscal surgery in the previous 6 weeks
* chemiotherapy, radioteherapy
* diabetes
* alchoolism, psichiatric disease,drug addiction
* coagulation disorders
* pregnancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Symptomatic and functional evaluation at 6 months by comparison of the KOOS score recorded between the two groups | 6 month
  Symptomatic and functional evaluation at 6 months by comparison of the KOOS score recorded between two groups (6±1 months) undergoing arthroscopic debridement ± injection of autologous microfragmented lipoaspirate tissue (Lipogems®).

SECONDARY OUTCOMES:
Radiological changes at 6 month recorded between the two groups | 6 month
  Evaluation of possible radiological changes pre-operative and after 6±1 months by means of MagneticResonanceImaging analysis.
Functional changes at 6 month recorded between the two groups | 6 month
  Symptomatic and functional evaluation at 6±1 months by means of Proms that inclued questionnaire about quality of life (SF-12, WOMAC)
Serum changes at 6 month recorded between the two groups | 6 month
  Changes in serum levels of biomarkers related to Osteoarthritis (collagen type II C-telopeptide(CTx-II),collagen type III N-propeptide( PIIINP)) will be evaluated (pre-intervention vs 6±1 months).

CONTACTS AND LOCATIONS:
Overall Officials: michele ulivi, Principal Investigator — IRCCS Istituto Ortopedico GaleazziMilano
Locations (2):
- Italy (2):
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Istituto Ortopedico Galeazzi, Milan